CLINICAL TRIAL: NCT06661551
Title: Does the Generation to Which the Operator Belongs Influence the Orthodontic Miniscrew Insertion Accuracy in Dynamic Computer-guided Surgery? a Randomized Clinical Prospective Study
Brief Title: Does the Generation to Which the Operator Belongs Influence the Orthodontic Miniscrew Insertion Accuracy in Dynamic Computer-guided Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Michele Cassetta, DDS, PhD, Full Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URomLS_5951
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Malocclusion; Malocclusion in Children; Malocclusion; Displaced or Missing Teeth
Keywords: Dynamic computer-guided surgery; navigation systems; TADs; generations; accuracy
MeSH Terms: conditions — Malocclusion; Anodontia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Generation X operator) (Experimental): Group A is going to be treated by operator number 1, an oral surgeon with more than 30 Years of experience, which belongs to "Generation X"
  Interventions: Procedure: Miniscrew insertion in dynamic-computer guided surgery
- Group B (Generation Y operator) (Experimental): Operator number 2 (MG) will treat Group B and is a dentist with 15 years of experience in oral surgery and belonged to "Generation Y".
  Interventions: Procedure: Miniscrew insertion in dynamic-computer guided surgery
- Group C (Generation Z operator) (Experimental): Group C will be treated by operator number 3 (DB), a final year dental student with no previous experience in oral surgery, that belonged to "Generation Z".
  Interventions: Procedure: Miniscrew insertion in dynamic-computer guided surgery

INTERVENTIONS:
Procedure: Miniscrew insertion in dynamic-computer guided surgery — The intervention more executed in the literature is by using static computer-guided systems (s-CAS) . However, the s-CAS has limitations, including the time and cost associated with guide production, furthermore, the guide's bulk prevents its use in patients with limited mouth opening, and reduced irrigation potentially leads to overheating and bone burns during implant placement. Additionally, the inability to adjust the surgical plan intraoperatively, the lack of real-time visualization during implant site preparation and implant insertion, and the requirement for specific surgical kits for each implant system present further challenges.
  Dynamic navigation systems offer several benefits as highlighted in the literature, including: real-time feedback of the position of surgical drill or implant, allowing intraoperative changes adjusting the implant position during the surgery, reduction of risk of injury to adjacent anatomical structures, promotion of accuracy in novices

SUMMARY:
The goal of this clinical trial is to access the miniscrew accuracy insertion via dynamic computer-guided systems, inserted by three different clinicians belonging to three different generations, in childern in late mixed dentition or permanent dentition that need for orthodontic treatment, with good oral hygiene and absence of acute infection in the oral cavity and good general healt. The main questions it aims to answer are:

* Are there statistically significant differences between accuracy parameters and generation to which the clinician belongs?
* Does exist a significant correlation between the deviation parameters and the number of surgeries, and between the duration of interventions and the number of surgeries? Researchers wirll compare the deviation parameters to see if there are statistically significant differences in terms of accuracy.

Participants will undergo a surgical procedure of placement of 2 orthodontic miniscrews in the palatal region, and then a post-operative CBCT to assess the accuracy and presence or absence of damage to adjacent structures

DETAILED DESCRIPTION:
This study will be conducted to evaluate intergenerational differences regarding orthodontic miniscrew placement accuracy in the palatine vault through dynamic computer-guided surgery. The secondary outcome will be to assess, for each operator, the correlation between the number of miniscrews inserted, i.e. surgeries, and the accuracy variables as well as the duration of interventions.

The clinical investigation will be conducted between December 2022 and September 2024, adhering to the ethical standards outlined in the seventh revision of the Declaration of Helsinki. Parents and guardians are going to be informed about the details of the study, including the benefits and potential risks, and provided written consent. The investigation is approved by the local ethics committee (no. 5951).

The eligibility criteria are: (1) children in late mixed dentition or permanent dentition, (2) need for orthodontic treatment, (3) good oral hygiene, (4) absence of acute infection in the oral cavity, (5) good general health. The exclusion criteria are as follows: (1) syndromic patients, (2) uncontrolled systemic disease.

Miniscrews will be placed by three different clinicians, belonging to three different generations and levels of experience in implant and orthodontic miniscrew placement in free-hand and static computer-guided surgery.

A block randomization sequence is going to be generated using the Sealed Envelope online tool (https://www.sealedenvelope.com) to allocate the subjects into three groups. The random allocation sequence generation, enrollment, and assignment of the participants to interventions will be done by an external researcher not involved in the research. The allocation ratio of the subjects will be balanced, based on the generation to which the researchers belong.

Group A is going to be treated by operator number 1, an oral surgeon with more than 30 Years of experience, which belongs to "Generation X"; operator number 2 (MG) will treat Group B and is a dentist with 15 years of experience in oral surgery and belonged to "Generation Y"; Group C will be treated by operator number 3 (DB), a final year dental student with no previous experience in oral surgery, that belonged to "Generation Z". However, all three were novices in the use of dynamic computer-guided surgical systems, and no pre-clinical training phase was done.

In order to achieve skeletal anchorage for orthodontic or orthopedic treatment, the miniscrews (BENEfit®, Benefit system; PSM Medical Solutions, Tuttlingen, Germany) will be inserted under local anesthesia, in the paramedian area of the hard palate at the level of the third palatine rugae, and to guarantee a minimally-invasive, flapless and pre-drilling free approach, the miniscrews will be inserted using the Navident dynamic navigation system (ClaroNav Technology Inc., Toronto, Canada), through a NSK iSD900 cordless battery screwdriver (Nakanishi INC., Tochigi, Japan).

The patients will undergo to optical scanning, using a Medit i700 intraoral scanner (Medit Corp., Seoul, South Korea) and CBCT imaging of the upper jaw, captured using a Scanora 3Dx cone-beam device (Soredex, Tuusula, Finland).

The resulting STL (Standard Triangulation Language) and DICOM (Digital Imaging and Communications in Medicine) files are going to be superimposed to precisely determine the insertion site, diameter, and length of the miniscrews to achieve bicortical anchorage.

To evaluate the accuracy of miniscrew placement and to detect any potential root injury, a postoperative CBCT scan was conducted immediately after each surgical procedure.

The preoperative and postoperative images were superimposed, through the use of EvaluNav software (ClaroNav Technology Inc., Toronto, Canada), employing coordinated automatically given by the software as previously described [3, 10, 26]. To assess the differences between the planned position and the actual placement of miniscrews, five deviation parameters will be analyzed: Entry-3D, Entry-2D, Apex-3D, Apex vertical (vertical deviation), Angular deviation (Figure 2) The duration of the surgeries will be calculated by an external researcher using the Navident Software (ClaroNav Technology Inc., Toronto, Canada) from the moment when the Navigation View appears to the end of the navigation phase.

The sample size was calculated based on a previous study using G*Power software (version 3.1.9.6; Heinrich-Heine-Universität Düsseldorf, Düsseldorf, Germany). The significance level was set at 0.05 and the power at 0.8. A total sample size of thirty-three os considered acceptable, with an actual power of 0.81.

To reduce the risk of statistical analysis bias, the operator variable will be coded, and a blinded statistician will perform the statistical analysis, using Excel (Microsoft, Redmond, Washington, USA) to create a database to allocate the subjects, and the statistical software package SPSS version 27.0 (IBM Corp., New York, USA).

Descriptive statistics analysis (including mean, minimum, maximum values, confidence interval at 95% and standard deviations) is going to be performed for each variable within each group.

Subsequently, the Shapiro-Wilk normality test will be conducted to assess the distribution of the data. For variables following a normal distribution, the ANOVA test will be employed; whereas, for variables exhibiting a non-normal distribution, a non-parametric test, namely the Kruskal-Wallis H test, is performed. In cases where the tests indicated statistically significant differences, post-hoc tests will be subsequently conducted. The Tukey test is going to be used for variables with a normal distribution, and the Dunn's for a non-normal distribution.

Furthermore, the Pearson Correlation will be utilized to analyze whether the number of surgeries influenced the deviation variables (Entry-3D, Entry-2D, Apex-3D, Apex Vertical, Angular deviation, duration of the intervention).

The level of significance was set at P ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Children in late mixed dentition or permanent dentition;
* Need for orthodontic treatment;
* Good oral hygiene;
* Absence of acute infection in the oral cavity;
* Good general health.

Exclusion Criteria:

* Syndromic patients;
* Uncontrolled systemic disease.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Miniscrew insertion accuracy assessment | Through study completion, and average of 1 year and a half
  The preoperative and postoperative DICOM images need to be superimposed, through the use of EvaluNav software (ClaroNav Technology Inc., Toronto, Canada), employing coordinated automatically given by the software. The software, to assess the differences between the planned position and the actual placement of miniscrews, will provide five deviation parameters: Entry-3D, Entry-2D, Apex-3D, Apex vertical (vertical deviation), Angular deviation.
  Entry 2D: deviation of the miniscrew platform in the x and y dimensions of space in an occlusal view; Entry 3D: deviation of the miniscrew platform in the three dimensions of space; Apex 3D: deviation of the miniscrew apex in the three dimensions of space; Apex vertical: deviation of miniscrew apex depth (z-axis), in millimeters (mm); Angle: angular deviation between the central axes of the planned position and the final position, in degrees (°).

SECONDARY OUTCOMES:
Correlation between the deviation parameters and the number of surgeries, and between the duration of interventions and the number of surgeries. | Through study completion, and average of 1 year and a half
  The Pearson Correlation will be utilized to analyze whether the number of surgeries influenced the deviation variables (Entry-3D, Entry-2D, Apex-3D, Apex Vertical, Angular deviation, duration of the intervention).

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Umberto I, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brilli D, Cauli I, Cassetta M. How palatal vault morphology and screw length influence the accuracy of dynamic computer-guided orthodontic miniscrew insertion. A prospective clinical study. J Dent. 2024 Jul;146:105093. doi: 10.1016/j.jdent.2024.105093. Epub 2024 May 22. PMID 38788916
- [Background] S. Bertoldo, D. Brilli, I. Cauli, M. Cassetta, Dynamic navigation for miniscrew insertion in the palatal vault: a pilot study, Dental Cadmos 7 (2024). https://doi.org/10.19256/d.cadmos.07.2024.06.
- [Derived] Brilli D, Giansanti M, Cassetta M. Does the operator's generational cohort influence the accuracy of orthodontic miniscrews insertion in the palatine vault in dynamic computer-guided surgery? A randomized prospective study. Oral Maxillofac Surg. 2025 Jun 10;29(1):120. doi: 10.1007/s10006-025-01414-7. PMID 40493264